CLINICAL TRIAL: NCT02425891
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled Study of Atezolizumab (Anti-PD-L1 Antibody) in Combination With Nab-Paclitaxel Compared With Placebo With Nab-Paclitaxel for Patients With Previously Untreated Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of Atezolizumab in Combination With Nab-Paclitaxel Compared With Placebo With Nab-Paclitaxel for Participants With Previously Untreated Metastatic Triple-Negative Breast Cancer (IMpassion130)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO29522; 2014-005490-37 (EudraCT Number)
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Atezolizumab Plus Nab-Paclitaxel (Experimental): Participants assigned to atezolizumab plus nab-paclitaxel received both agents until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PDL1 antibody; Drug: Nab-Paclitaxel
- Placebo Plus Nab-Paclitaxel (Placebo Comparator): Participants assigned to placebo plus nab-paclitaxel received both agents until disease progression or unacceptable toxicity.
  Interventions: Drug: Nab-Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PDL1 antibody — Atezolizumab at a fixed dose of 840 milligrams via intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Other Names: Tecentriq, MPDL3280A
  Arms: Atezolizumab Plus Nab-Paclitaxel
Drug: Nab-Paclitaxel — Nab-Paclitaxel at a starting dose of 100 milligrams per square meter via IV infusion on Days 1, 8, and 15 of each 28-day cycle. Nab-Paclitaxel was administered for a target of at least 6 cycles, with no maximum in the absence of disease progression or unacceptable toxicity.
  Other Names: Abraxane®
Drug: Placebo — Placebo administered via IV infusion on Days 1 and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
  Arms: Placebo Plus Nab-Paclitaxel

SUMMARY:
This multicenter, randomized, double-blind study evaluated the efficacy, safety, and pharmacokinetics of atezolizumab (MPDL3280A) administered with nab-paclitaxel compared with placebo in combination with nab-paclitaxel in participants with locally advanced or metastatic triple-negative breast cancer (TNBC) who have not received prior systemic therapy for metastatic breast cancer (mBC). The safety of single-agent nab-paclitaxel has been determined in previous studies of participants with mBC and the safety data to date suggest that atezolizumab can be safely combined with standard chemotherapy agents.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced, histologically documented TNBC characterized by absence of human epidermal growth factor 2 (HER2), estrogen receptor (ER), and progesterone receptor (PR) expression
* No prior chemotherapy or targeted systemic therapy for inoperable locally advanced or metastatic TNBC
* Eligible for taxane monotherapy (i.e., absence of rapid clinical progression, life-threatening visceral metastases, or the need for rapid symptom and/or disease control)
* A representative formalin-fixed, paraffin-embedded tumor specimen in paraffin blocks, or at least 20 unstained slides with an associated pathology report documenting ER, PR, and HER2 negativity. Participants with fewer than 20 unstained slides available at baseline, and not fewer than 12 unstained slides will be eligible upon discussion with Medical Monitor
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Measurable disease as defined by RECIST v1.1
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases
* Leptomeningeal disease
* Pregnancy or lactation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Receipt of a live, attenuated vaccine within 4 weeks prior to randomization, during treatment, or within 5 months following the last dose of atezolizumab/placebo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (247):
- United States (49):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente of Northern California, Oakland, California
  - Emad Ibrahim, Md, Inc, Redlands, California
  - Univ of Calif, San Francisco; Breast Cancer Center, San Francisco, California
  - Kaiser Permanente - San Marcos, San Marcos, California
  - Cancer Research Collaboration, Inc., Santa Ana, California
  - Stanford Univ School of Med; Oncology, Stanford, California
  - Kaiser Permanente Of Colorado, Aurora, Colorado
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Stamford Hospital; BCC, MOHR, Stamford, Connecticut
  - MedStar Georgetown University Hospital (Lombardi Comprehensive Cancer Center), Washington D.C., District of Columbia
  - Florida Cancer Specialists - SCRI; Pharmacy, Fort Myers, Florida
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - The Mount Siani Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Rush University Medical Center - Chicago, Chicago, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Maryland Oncology Hematology, Rochville, Maryland
  - Barbara Ann Karmanos Cancer Institute; Oncology, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Health Midwest Ventures Group, Inc d/b/a HCA MidAmerica Division, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New Hampshire Hematology Oncology, Manchester, New Hampshire
  - The Valley Hospital, Ridgewood, New Jersey
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Onc/Hem Care Clin Trials LLC, Cincinnati, Ohio
  - The Mark H. Zangmeister Ctr; Mid Ohio Onc/Hem Inc., Columbus, Ohio
  - Kaiser Perm NW - Rheuma, Portland, Oregon
  - Providence Cancer Center, Portland, Oregon
  - St. Luke's Cancer Care Associates, Bethlehem, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Greenville Health System (GHS) Cancer Institute, Greenville, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - West Clinic, Germantown, Tennessee
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Texas Oncology- El Paso Cancer Treatment Center Gateway, El Paso, Texas
  - The Methodist Cancer Center, Houston, Texas
  - University of Texas;M.D. Anderson Cancer Center, Houston, Texas
  - Inova Medical Group, Fairfax, Virginia
  - Cancer Care Northwest, Spokane, Washington
- Argentina (3):
  - Centro de Oncologia e Investigacion Buenos Aires (COIBA), Buenos Aires
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
- Australia (8):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Nepean Cancer Care Centre, Sydney, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Princess Alexandra Hospital; Division of Cancer Services, Woolloongabba, Queensland
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - St John of God Hospital; Bendat Cancer Centre, Subiaco, Western Australia
- Austria (4):
  - Lkh-Univ. Klinikum Graz; Klinik Für Innere Medizin I, Graz
  - Ordensklinikum Linz Barmherzige Schwestern; Abt. fur Innere Medizin 1, Linz
  - A.Ö. Lhk; Ii. Medizinische Abt. Mit Schwerpunkt Gaströnter. & Onkologie, Steyr
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I, Vienna
- Belgium (6):
  - Institut Jules Bordet, Anderlecht
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Notre Dame, Charleroi
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
  - Sint Augustinus Wilrijk, Wilrijk
- Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (10):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital Perola Byington, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
- Canada (11):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - BC Cancer - Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Chile (2):
  - Centro de Cancer Pontificie Universidad Catolica de Chile, Santiago
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
- Colombia (2):
  - Clinica del Country, Bogotá
  - Oncomedica S.A., Montería
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- Czechia (3):
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
  - Fakultni nemocnice v Motole, Prague
- Estonia (2):
  - North Estonia Medical Centre Foundation; Oncology Centre, Tallinn
  - Tartu Uni Hospital; Hematology - Oncology Clinic, Tartu
- Tampere University Hospital; Dept of Oncology, Tampere, Finland
- France (12):
  - Ico - Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Hopital Jean Minjoz, Besançon
  - HOPITAL MICHALLON - CENTRE HOSPITALIER UNIVERSITAIRE DE GRENOBLE, Service d'oncologie Médicale, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut régional du Cancer Montpellier, Montpellier
  - Clinique Catherine de Sienne, Nantes
  - Institut Curie, Paris
  - Hopital La Pitie Salpetriere, Paris
  - Institut De Cancerologie De L'Ouest; Medical Oncology, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
- Germany (20):
  - Ambulantes Tumorzentrum Spandau; Dres. Benno Mohr und Uwe Peters, Berlin
  - St. Elisabeth-Krankenhaus; Brustzentrum, Cologne
  - St. Johannes Hospital; Abt. für Hämatologie und Onkologie, Dortmund
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - Uniklinik Essen; Gynäkologie, Essen
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg GmbH, Georgsmarienhütte
  - Universitätsklinikum Halle (Saale); Universitätsklinik Und Poliklinik Für Gynäkologie, Halle
  - Universitätsklinikum Hamburg-Eppendorf; Frauenklinik, Hamburg
  - Facharztzentrum Eppendorf, Studien GbR, Hamburg
  - Universitatsklinik Heidelberg; Universitätshautklinik und Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Praxis Köppler, Heymann, Weide, Thomalla; Fä Für Innere Medizin, Koblenz
  - Universitätsklinikum Schleswig-Holstein; Campus Lübeck, Lübeck
  - Klinikum rechts der Isar der TU München; Klinik und Poliklinik für Frauenheilkunde, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - MVZ Nordhausen gGmbH, Praxis Dr. Grafe, Nordhausen
  - Oncologianova GmbH - Gesellschaft für Innovationen in der Onkologie, Recklinghausen
  - Mutterhaus der Borromäerinnen gGmbH, Abteilung Hämatologie-Onkologie, Trier
  - Dres. Helmut Forstbauer, Carsten Ziske und Kollegen; Onkologische Schwerpunktpraxis, Troisdorf
  - Universitätsklinik Tübingen; Frauenklinik & Poliklinik, Tübingen
- Greece (5):
  - Anticancer Hospital Ag Savas; 1St Dept of Internal Medicine, Athens
  - IASO General Hospital of Athens, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Patras Medical Oncology, Pátrai
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
- Grupo Angeles, Guatemala City, Guatemala
- Queen Mary Hospital; Dept of Medicine, Hong Kong, Hong Kong
- Hungary (3):
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Italy (2):
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Irccs Istituto Europeo Di Oncologia (IEO); Ricerca Di Senologia Medica, Milan, Lombardy
- Japan (27):
  - Aichi Cancer Center Hospital, Aichi
  - Fukushima Medical University Hospital, Fukushima
  - Gunma Prefectural Cancer Center, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - Sagara Hospital, Kagoshima
  - St. Marianna University Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Tohoku University Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Naha-nishi Clinic, Okinawa
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Latvia (2):
  - Daugavpils Regional Hospital, Daugavpils
  - Riga East Clinical University Hospital Latvian Oncology Centre, Riga
- Mexico (5):
  - Centro Medico Dalinde, Mexico City, Mexico CITY (federal District)
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Instituto Estatal de Cancerologia Colima, Colima
  - Iem-Fucam, D.F.
  - Consultorio de Medicina Especializada; Dentro de Condominio San Francisco, Mexico City
- Norway (3):
  - Helse Bergen HF Haukeland universitetssjukehus kreftavdelingen poliklinikk, Bergen
  - Sørlandet Sykehus Kristiansand, Kristiansand
  - Stavanger Universitetssykehus, Helse Stavanger HF, Stavanger
- Centro Oncológico de Panamá, Panama City, Panama
- Poland (6):
  - Centrum Onkologii w Bydgoszczy; Oddzial Kliniczny Onkologii, Bydgoszcz
  - Szpitale Wojewodzkie w Gdyni Sp. z o.o., Gdynia
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Centrum Onkologii Ziemi LUBELSKIEJ im. Sw Jana z Dukli, I oddz. Chemioterapii, Lublin
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad; Klinika Nowtw.Piersi i Chir.Rekonstr, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Oncomed SRL, Timișoara, Romania
- Russia (7):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Main Military Clinical Hospital named after N.N. Burdenko, Moscow, Moscow Oblast
  - Blokhin Cancer Research Center; Combined Treatment, Moskva, Moscow Oblast
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Instituto Valenciano Oncologia; Oncologia Medica, Valencia
- Sweden (2):
  - Sodersjukhuset; Onkologkliniken, Stockholm
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Switzerland (3):
  - Universitaetsspital Basel; Onkologie, Basel
  - Kantonsspital St.Gallen Brustzentrum/Chirurgie; Brustzentrum, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- Taiwan (4):
  - Kaohsiung Medical Uni Chung-Ho Hospital; Dept of Surgery, Kaohsiung City
  - China Medical University Hospital; Surgery, Taichung
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; General Surgery, Taipei
- Thailand (3):
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- Turkey (Türkiye) (5):
  - Cukurova Uni Faculty of Medicine; Medical Oncology, Adana
  - Istanbul University Cerrahpasa Medical Faculty; Radiation Oncology Department, Istanbul
  - Medipol University MF; Oncology Department, Istanbul
  - Ege Uni Medical Faculty Hospital; Oncology Dept, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- Ukraine (4):
  - Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - Kyiv City Clinical Oncological Center, Kyiv
  - Treatment and Prevention Institution Volyn Regional Oncology Dispensary, Lutsk
  - Lviv State Oncology Regional Treatment and Diagnostic Centre, Lviv
- United Kingdom (10):
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital; Clinical Oncology, Edinburgh
  - St Bartholomew's Hospital, London
  - Guys ST Thomas Hospital, London
  - Royal Marsden Hospital - London, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Derriford Hospital, Plymouth
  - Royal Preston Hosptial, Preston
  - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Li M, Yang B. Prognostic Value of NUSAP1 and Its Correlation with Immune Infiltrates in Human Breast Cancer. Crit Rev Eukaryot Gene Expr. 2022;32(3):45-60. doi: 10.1615/CritRevEukaryotGeneExpr.2021040248. PMID 35695609
- [Derived] Wang H, Ma H, Sove RJ, Emens LA, Popel AS. Quantitative systems pharmacology model predictions for efficacy of atezolizumab and nab-paclitaxel in triple-negative breast cancer. J Immunother Cancer. 2021 Feb;9(2):e002100. doi: 10.1136/jitc-2020-002100. PMID 33579739
- [Derived] Adams S, Dieras V, Barrios CH, Winer EP, Schneeweiss A, Iwata H, Loi S, Patel S, Henschel V, Chui SY, Rugo HS, Emens LA, Schmid P. Patient-reported outcomes from the phase III IMpassion130 trial of atezolizumab plus nab-paclitaxel in metastatic triple-negative breast cancer. Ann Oncol. 2020 May;31(5):582-589. doi: 10.1016/j.annonc.2020.02.003. Epub 2020 Feb 20. PMID 32178964
- [Derived] Schmid P, Rugo HS, Adams S, Schneeweiss A, Barrios CH, Iwata H, Dieras V, Henschel V, Molinero L, Chui SY, Maiya V, Husain A, Winer EP, Loi S, Emens LA; IMpassion130 Investigators. Atezolizumab plus nab-paclitaxel as first-line treatment for unresectable, locally advanced or metastatic triple-negative breast cancer (IMpassion130): updated efficacy results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Jan;21(1):44-59. doi: 10.1016/S1470-2045(19)30689-8. Epub 2019 Nov 27. PMID 31786121
- [Derived] Schmid P, Adams S, Rugo HS, Schneeweiss A, Barrios CH, Iwata H, Dieras V, Hegg R, Im SA, Shaw Wright G, Henschel V, Molinero L, Chui SY, Funke R, Husain A, Winer EP, Loi S, Emens LA; IMpassion130 Trial Investigators. Atezolizumab and Nab-Paclitaxel in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2018 Nov 29;379(22):2108-2121. doi: 10.1056/NEJMoa1809615. Epub 2018 Oct 20. PMID 30345906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The observation of Overall Survival events was complete. Participants still on treatment were handed over to follow-up programs or studies. The study status is "Completed" but some participants discontinued the study because the Sponsor terminated it after it reached the "Completed" state.
Period: Overall Study
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Started | 451 | 451
Completed | 0 | 0
Not Completed | 451 | 451
Not completed — Death | 333 | 314
Not completed — Lost to Follow-up | 4 | 6
Not completed — Non-Compliance | 1 | 1
Not completed — Accidentally randomized screen failure participant | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Study Terminated By Sponsor | 85 | 95
Not completed — Withdrawal by Subject | 27 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel | Total
Number analyzed (Participants) | 451 | 451 | 902
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (12.1) | 54.3 (12.3) | 54.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 450 | 449 | 899
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 60 | 143
  Not Hispanic or Latino | 340 | 368 | 708
  Unknown or Not Reported | 28 | 23 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 17 | 40
  Asian | 76 | 85 | 161
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 32 | 26 | 58
  White | 301 | 308 | 609
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) in All Randomized Participants
Description: PFS was defined as the time from randomization to the occurrence of disease progression, as determined by investigators from tumor assessments per RECIST v1.1, or death from any cause, whichever occurred first.
Time Frame: Baseline up to approximately 34 months
Population: The ITT population is defined as all randomized patients, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 451 | 451
Months | 5.49 [5.32 to 5.59] | 7.16 [5.59 to 7.46]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.0025, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.69 to 0.92]

2. Primary Outcome: PFS According to RECIST v1.1 in Participants With Detectable Programmed Death-Ligand 1 (PD-L1)
Description: as for outcome 1
Time Frame: Baseline up to approximately 34 months
Population: The PD-L1-selected subpopulation is defined as patients in the ITT population whose PD-L1 status is IC1/2/3 at the time of randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 184 | 185
Months | 4.96 [3.81 to 5.55] | 7.46 [6.70 to 9.23]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p < .0001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.49 to 0.78]

3. Primary Outcome: Overall Survival (OS) in All Randomized Participants
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline until death due to any cause (up to approximately 58 months)
Population: The ITT population is defined as all randomized patients, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 451 | 451
Months | 18.73 [16.85 to 20.76] | 21.03 [19.02 to 23.36]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.0770, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.75 to 1.02]

4. Primary Outcome: OS in Participants With Detectable PD-L1
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline until death due to any cause (up to approximately 58 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 184 | 185
Months | 17.91 [13.63 to 20.30] | 25.43 [19.55 to 30.69]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.0016, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.53 to 0.86]

5. Secondary Outcome: Percentage of Participants With an Objective Response of Complete Response (CR) or Partial Response (PR) According to RECIST v1.1 in All Randomized Participants
Description: An objective response was defined for participants with measurable disease at baseline as either a partial response (PR) or a complete response (CR) using RECIST v1.1.
Time Frame: Baseline up to approximately 34 months
Population: The ORR-evaluable population is defined as patients in the ITT population with measurable disease at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 449 | 450
Percentage of Participants | 45.9 | 56.0
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.0021, Cochran-Mantel-Haenszel; Difference in Overall Response Rates = 10.12, 95% CI 2-sided [3.40 to 16.84]

6. Secondary Outcome: Percentage of Participants With an Objective Response of CR or PR According to RECIST v1.1 in Participants With Detectable PD-L1
Description: as for outcome 5
Time Frame: Baseline up to approximately 34 months
Population: The PD-L1-ORR-evaluable population is defined as patients in the PD-L1-selected subpopulation with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 183 | 185
Percentage of participants | 42.6 | 58.9
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.0016, Cochran-Mantel-Haenszel; Difference in Overall Response Rates = 16.30, 95% CI 2-sided [5.67 to 26.92]

7. Secondary Outcome: Duration of Response (DOR) According to RECIST v1.1 in All Randomized Participants
Description: DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response (CR or PR) to the date of disease progression per RECIST v1.1 or death from any cause, whichever occurred first.
Time Frame: Baseline up to approximately 34 months
Population: The duration of response (DOR)-evaluable population is defined as patients with an objective response.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 206 | 252
Months | 5.62 [5.52 to 6.93] | 7.39 [6.90 to 9.00]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Unstratified Analysis; p = 0.0285, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.63 to 0.98]

8. Secondary Outcome: DOR Acccording to RECIST v1.1 in Participants With Detectable PD-L1
Description: as for outcome 7
Time Frame: Baseline up to approximately 34 months
Population: The duration of response (DOR)-evaluable population is defined as patients with an objective response.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 78 | 109
Months | 5.49 [3.71 to 7.13] | 8.48 [7.33 to 9.66]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Unstratified Analysis; p = 0.0047, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.43 to 0.86]

9. Secondary Outcome: Time to Deterioration (TTD) in Global Health Status/Health Related Quality of Life According to European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) v3.0 in All Randomized Participants
Description: Deterioration in GHS/HRQoL (Items 29, 30 of the EORTC QLQ C30) was defined by the following two criteria: 1. The time from randomization to the first time the participant's GHS/HRQoL scale score showed a >=10-point decrease from the baseline scale score. A 10-point change was defined as the minimally important difference (MID). 2. The score decrease of >= 10-points from baseline was held for at least two consecutive cycles, or an initial score decrease of >= 10-points was followed by death or treatment discontinuation within 3 weeks from the last assessment.
Time Frame: Baseline up to approximately 58 months
Population: The patient-reported outcome (PRO)-evaluable population is defined as patients in the ITT population with a baseline and ≥1 post-baseline PRO assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 400 | 406
Months | 7.98 [5.65 to 11.10] | 8.18 [6.01 to 10.94]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.8078, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.81 to 1.18]

10. Secondary Outcome: TTD in Global Health Status/Health Related Quality of Life According to EORTC QLQ-C30 v3.0 in Participants With Detectable PD-L1
Description: Deterioration in GHS/HRQoL (Items 29, 30 of the EORTC QLQ C30) was defined by the following two criteria: 1. The time from randomization to the first time the participants's GHS/HRQoL scale score showed a >=10-point decrease from the baseline scale score. A 10-point change was defined as the minimally important difference (MID). 2. The score decrease of >= 10-points from baseline was held for at least two consecutive cycles, or an initial score decrease of >= 10-points was followed by death or treatment discontinuation within 3 weeks from the last assessment.
Time Frame: Baseline up to approximately 58 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 160 | 167
Months | 6.41 [4.57 to 11.24] | 7.56 [4.99 to 12.12]
Statistical Analysis 1: Comparison: Placebo Plus Nab-Paclitaxel vs Atezolizumab Plus Nab-Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.8879, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.73 to 1.31]

11. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: Percentage of participants with at least one adverse event.
Time Frame: Baseline up to to the data cutoff date: 31 August 2021 (up to approximately 74 months)
Population: The safety-evaluable population is defined as participants who received any amount of any study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab Plus Nab-Paclitaxel | Placebo Plus Nab-Paclitaxel
Number analyzed (Participants) | 460 | 430
Percentage of participants | 99.3 | 97.9

12. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) Against Atezolizumab
Description: Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) Against Atezolizumab
Time Frame: Baseline up to approximately 53 months
Population: The anti-drug antibodies (ADA)-evaluable population is defined as all patients treated with atezolizumab who have at least one post-baseline ADA result.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 434
Percentage of participants
  Baseline Prevalence of ADAs | 1.6
  Incidence of Treatment Emergent ADAs | 13.1

13. Secondary Outcome: Maximum Serum Concentration (Cmax) for Atezolizumab
Description: Maximum serum concentration for atezolizumab.
Time Frame: Cycle 1 Day 1 (Cycle = 28 days)
Population: The pharmacokinetic (PK)-evaluable population is defined as all patients who received any dose of study medication and who have at least one post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 407
µg/mL | 329 (98.9)

14. Secondary Outcome: Minimum Serum Concentration (Cmin) for Atezolizumab
Description: Minimum serum concentration for atezolizumab.
Time Frame: Day 27 of Cycle 1, 2, 3, and 7 (Cycle = 28 days)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 420
µg/mL
  Cycle 1 Day 27 | 145 (52.6)
  Cycle 2 Day 27: number analyzed (Participants) | 373
  Cycle 2 Day 27 | 215 (78.3)
  Cycle 3 Day 27: number analyzed (Participants) | 343
  Cycle 3 Day 27 | 245 (90.3)
  Cycle 7 Day 27: number analyzed (Participants) | 188
  Cycle 7 Day 27 | 274 (111)

15. Secondary Outcome: Plasma Concentrations of Total Paclitaxel
Description: Plasma Concentrations of Total Paclitaxel
Time Frame: Pre-dose (Hour 0) on Cycle 1 Day 1, pre-dose (Hour 0), 5-10 minutes before end of nab-paclitaxel infusion, 1 hour after end of nab-paclitaxel infusion (infusion duration = 30 minutes) on Cycle 3 Day 1 (Cycle = 28 days)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo Plus Nab-Paclitaxel | Atezolizumab Plus Nab-Paclitaxel
Number analyzed (Participants) | 321 | 436
ng/mL
  C1D1/Predose | NA (NA) — Cycle 1 predose is before study drug treatment. | NA (NA) — Cycle 1 predose is before study drug treatment.
  C3D1/Predose: number analyzed (Participants) | 310 | 351
  C3D1/Predose | NA (NA) — Below the level of detection as expected given the half-life of 13-27 hours per abraxane product label. | NA (NA) — Below the level of detection as expected given the half-life of 13-27 hours per abraxane product label.
  C3D1/ Before End of Infusion: number analyzed (Participants) | 255 | 298
  C3D1/ Before End of Infusion | 2970 (2300) | 3080 (2050)
  C3D1/Postdose Paclit: number analyzed (Participants) | 221 | 280
  C3D1/Postdose Paclit | 370 (244) | 400 (275)

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 31 August 2021 (up to approximately 74 months)
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any study drug. In placebo+nab-paclitaxel arm, 6 participants received atezolizumab in error & 9 participants crossed over from placebo+nab-paclitaxel arm to atezolizumab+nab-paclitaxel arm.
Groups:
- Placebo (q2w) + Nab-Paclitaxel: Participants assigned to placebo plus nab-paclitaxel received both agents until disease progression or unacceptable toxicity.
- Atezolizumab (q2w) + Nab-Paclitaxel: Participants assigned to atezolizumab plus nab-paclitaxel received both agents until disease progression or unacceptable toxicity.
Arm/Group | Placebo (q2w) + Nab-Paclitaxel | Atezolizumab (q2w) + Nab-Paclitaxel
All-Cause Mortality (participants affected / at risk) | 333/451 | 314/451
Serious Adverse Events (participants affected / at risk) | 80/430 | 110/460
Other Adverse Events (participants affected / at risk) | 414/430 | 450/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (q2w) + Nab-Paclitaxel (N=430) | Atezolizumab (q2w) + Nab-Paclitaxel (N=460)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (2) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ADDISON'S DISEASE (Endocrine disorders) | 0 (0) | 1 (1)
ADRENOCORTICAL INSUFFICIENCY ACUTE (Endocrine disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
HYPOPHYSITIS (Endocrine disorders) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 1 (1) | 0 (0)
KERATITIS (Eye disorders) | 0 (0) | 1 (1)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 2 (4)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 4 (5) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL TOXICITY (Gastrointestinal disorders) | 0 (0) | 1 (1)
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 2 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)
ASTHENIA (General disorders) | 1 (3) | 0 (0)
CATHETER SITE PAIN (General disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 2 (2)
ILL-DEFINED DISORDER (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 5 (5)
AUTOIMMUNE CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTOCHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 2 (2)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
SYSTEMIC IMMUNE ACTIVATION (Immune system disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (3) | 5 (5)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 2 (2)
ERYSIPELAS (Infections and infestations) | 2 (2) | 2 (4)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 (1) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MASTITIS (Infections and infestations) | 1 (1) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 12 (14)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (3)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 5 (5)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LIMB DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL THROMBOSIS (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
EMBOLIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
IIIRD NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
DEVICE BREAKAGE (Product Issues) | 0 (0) | 1 (1)
THROMBOSIS IN DEVICE (Product Issues) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LICHEN PLANUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1)
EMBOLISM (Vascular disorders) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 2 (2) | 1 (1)
PERIPHERAL EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BELL'S PALSY (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (q2w) + Nab-Paclitaxel (N=430) | Atezolizumab (q2w) + Nab-Paclitaxel (N=460)
ANAEMIA (Blood and lymphatic system disorders) | 115 (186) | 129 (221)
LEUKOPENIA (Blood and lymphatic system disorders) | 23 (50) | 30 (68)
NEUTROPENIA (Blood and lymphatic system disorders) | 66 (176) | 101 (238)
HYPOTHYROIDISM (Endocrine disorders) | 15 (15) | 67 (80)
DRY EYE (Eye disorders) | 15 (15) | 31 (33)
LACRIMATION INCREASED (Eye disorders) | 33 (33) | 28 (28)
ABDOMINAL PAIN (Gastrointestinal disorders) | 53 (63) | 53 (59)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 25 (26) | 29 (35)
CONSTIPATION (Gastrointestinal disorders) | 108 (132) | 115 (140)
DIARRHOEA (Gastrointestinal disorders) | 146 (212) | 151 (307)
DRY MOUTH (Gastrointestinal disorders) | 16 (17) | 39 (39)
DYSPEPSIA (Gastrointestinal disorders) | 31 (38) | 30 (34)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 12 (13) | 24 (26)
NAUSEA (Gastrointestinal disorders) | 164 (244) | 213 (338)
STOMATITIS (Gastrointestinal disorders) | 20 (24) | 49 (66)
VOMITING (Gastrointestinal disorders) | 73 (98) | 92 (141)
ASTHENIA (General disorders) | 51 (75) | 60 (80)
CHEST PAIN (General disorders) | 20 (22) | 33 (36)
CHILLS (General disorders) | 23 (26) | 42 (58)
FATIGUE (General disorders) | 194 (238) | 216 (264)
INFLUENZA LIKE ILLNESS (General disorders) | 11 (12) | 29 (35)
MUCOSAL INFLAMMATION (General disorders) | 16 (18) | 29 (38)
OEDEMA PERIPHERAL (General disorders) | 66 (86) | 73 (94)
PYREXIA (General disorders) | 45 (72) | 89 (145)
NASOPHARYNGITIS (Infections and infestations) | 36 (42) | 52 (80)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 38 (49) | 55 (84)
URINARY TRACT INFECTION (Infections and infestations) | 42 (60) | 57 (86)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 37 (38) | 53 (100)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 42 (48) | 49 (80)
NEUTROPHIL COUNT DECREASED (Investigations) | 49 (101) | 57 (163)
WEIGHT DECREASED (Investigations) | 26 (28) | 22 (26)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 21 (37) | 39 (89)
DECREASED APPETITE (Metabolism and nutrition disorders) | 80 (86) | 92 (117)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 10 (11) | 25 (33)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 9 (10) | 29 (45)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 11 (16) | 26 (62)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 88 (120) | 104 (174)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 59 (69) | 74 (106)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 11 (13) | 24 (28)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (5) | 25 (31)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 18 (20) | 25 (28)
MYALGIA (Musculoskeletal and connective tissue disorders) | 67 (86) | 72 (84)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 41 (53) | 56 (79)
DIZZINESS (Nervous system disorders) | 43 (49) | 69 (87)
DYSGEUSIA (Nervous system disorders) | 44 (50) | 52 (59)
HEADACHE (Nervous system disorders) | 92 (125) | 116 (172)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 97 (120) | 100 (138)
PARAESTHESIA (Nervous system disorders) | 29 (32) | 34 (44)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 52 (62) | 74 (90)
DEPRESSION (Psychiatric disorders) | 22 (22) | 18 (19)
INSOMNIA (Psychiatric disorders) | 52 (54) | 54 (59)
BREAST PAIN (Reproductive system and breast disorders) | 21 (22) | 31 (43)
COUGH (Respiratory, thoracic and mediastinal disorders) | 80 (116) | 127 (171)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 60 (68) | 70 (90)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 39 (43) | 36 (49)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 30 (37)
ALOPECIA (Skin and subcutaneous tissue disorders) | 247 (249) | 263 (272)
DRY SKIN (Skin and subcutaneous tissue disorders) | 25 (27) | 42 (45)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 30 (31) | 38 (39)
PRURITUS (Skin and subcutaneous tissue disorders) | 45 (53) | 73 (93)
RASH (Skin and subcutaneous tissue disorders) | 71 (96) | 84 (115)
HOT FLUSH (Vascular disorders) | 32 (35) | 30 (34)
HYPERTENSION (Vascular disorders) | 21 (32) | 25 (37)
LYMPHOEDEMA (Vascular disorders) | 30 (31) | 30 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT02425891/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT02425891/SAP_001.pdf